CLINICAL TRIAL: NCT05825469
Title: Development and Usability Testing of Nutrition Algorithms for Cancer Health Outcomes (NACHO) and Quality of Life During Cancer Treatment
Brief Title: Development and Testing of Nutritional Algorithms (NACHO)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Cancer Nutrition Consortium Inc. (Unknown)
Responsible Party: Principal Investigator, Marilyn Hammer, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-637
Record Dates: First submitted 2023-02-27; First posted 2023-04-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Nutrition Poor; Nutritional Deficiency; Quality of Life
Keywords: Poor Nutrition; Nutritional Deficiency; Quality of Life
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Algorithm (NACHO) (Experimental): Study procedures will be conducted as follows:
  * Development of nutrition algorithm by dietitian panel participants with oncology clinician consultation via convened group meetings.
  * Refinement of draft algorithms through feedback from participants and Family Advisory Council (PFAC) members.
  * Baseline questionnaires for participants.
  * Semi-structured interviews and/or focus groups with participants to evaluate algorithm usability and acceptability.
  * Participant questionnaires.
  Interventions: Behavioral: Nutrition Algorithm

INTERVENTIONS:
Behavioral: Nutrition Algorithm — A technology-based platform for a person-centered nutrition program, providing suggested foods and recipes from dietitians.
  Other Names: Nutrition Algorithm for Cancer Health Outcomes (NACHO) Program

SUMMARY:
The goal of this research study is to develop a nutrition algorithm to optimize nutritional status and improve quality of life during for participants who are completing or have completed cancer treatment.

The name of the intervention used in this research study is:

Nutrition Algorithm for Cancer Health Outcomes (NACHO) (a technology-based platform that houses the algorithms for the person-centered nutrition program)

DETAILED DESCRIPTION:
This is a longitudinal, mixed-methods, pilot descriptive study to develop a nutrition algorithm for cancer patients based on the Cancer Nutrition Consortium (CNC) study findings and refined through a dietitian panel participants and from feedback from participants and Family Advisory Council (PFAC) members.

Research study procedures include screening for eligibility, interviews and/or focus groups, dietitian panel meetings, and surveys.

Participation in this study is expected to last about 12 months.

It is expected about 130 people will participate in this research study.

ELIGIBILITY:
Inclusion Criteria for Dietitians/Oncology clinicians - Have worked with at least 3 patients at the study site who had nutritional challenges

Inclusion Criteria for Patient and Family Advisory Council (PFAC) participants

* Current member of adult PFAC
* > 18 years old

Inclusion Criteria for Patient participants

* > 18 years old
* Able to speak and read English
* Completed primary treatment (aim 2b) or actively undergoing treatment (aim 2b and aim 3, exploratory)
* Access to a device (e.g., computer, tablet, smartphone) through which they can receive and engage with a REDCap link

Exclusion Criteria for Patient Participants

• Provider does not recommend

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Nutrition Algorithm | 12 months
  Primary study endpoint is development of a nutrition algorithm using the Cancer Nutrition Consortium (CNC) study findings and iteratively refine through an expert Dana-Farber Cancer Institute dietary panel along with consultations from oncology clinicians as needed and feedback from a panel of 4-6 Patient and Family Advisory Council (PFAC) members. Specific to data analyses, chi square, fisher's exact tests, and linear regression will be used to evaluate characteristics associated with changes in taste and different food preferences over time. Findings will inform the development of the algorithms.

SECONDARY OUTCOMES:
Acceptability of Nutrition Algorithm for Cancer Health Outcomes (NACHO) Program | Up to 8 months
  Assessed using the System Usability Scale (SUS), a 10-item instrument with scores that range from 0-100 with higher scores representing greater usability. Acceptability is defined as a SUS score of >70.
Participant Satisfaction | Up to 8 months
  Assessed using the Acceptability e-Scale (AES), a six-item scale that measures how easy, enjoyable, understandable, and helpful the intervention is. Total scores range from 6-30 with higher scores representing greater acceptability. Acceptability is defined as a AES score of >24.
Panel member characteristics (Aims 1a, 1b, 2a, 2b) - Age | Up to 12 months
  Age group (i.e., 18-29, 30-39, 40-49, 50-59, 60-69, 70-79, 80+)
Panel member characteristics (Aims 1a, 1b, 2a, 2b) - Gender identity | Up to 12 months
  Gender identity (i.e., female, male, other____, prefer not to answer)
Panel member characteristics (Aims 1a, 1b, 2a, 2b) - Ethnicity | Up to 12 months
  Ethnicity (i.e., Hispanic/Latinx / non-Hispanic/non-Latinx, prefer not to answer)
Panel member characteristics (Aims 1a, 1b, 2a, 2b) - Race | Up to 12 months
  Race (i.e., Black, Caucasian, Asian, Native American, Pacific Islander, Alaska Native, multiracial, prefer not to answer)
Panel member characteristics (Aims 1a, 1b, 2a, 2b) - Position | Up to 12 months
  Position / role and years in position (non-patient panel members only) (fill in)
Characteristics of the cohort of 100 patients (Aim 3) - Age | Up to 12 months
  Age group (i.e., 18-29, 30-39, 40-49, 50-59, 60-69, 70-79, 80+)
Characteristics of the cohort of 100 patients (Aim 3) - Gender identity | Up to 12 months
  Gender identity (i.e., female, male, other____, prefer not to answer)
Characteristics of the cohort of 100 patients (Aim 3) - ethnicity | Up to 12 months
  Ethnicity (i.e., Hispanic/Latinx / non-Hispanic/non-Latinx, prefer not to answer)
Characteristics of the cohort of 100 patients (Aim 3) - race | Up to 12 months
  Race (i.e., Black, Caucasian, Asian, Native American, Pacific Islander, Alaska Native, multiracial, prefer not to answer)
Characteristics of the cohort of 100 patients (Aim 3) - BMI | Up to 12 months
  Body mass index will will be calculated from weight in pounds and height in inches using the formula: weight (lb) / [height (in)]squared x 703
Characteristics of the cohort of 100 patients (Aim 3) - Comorbidities | Up to 12 months
  Comorbidities: Number of comorbidities (e.g., heart disease, diabetes) will be abstracted from electronic health records
Global Health | Up to 12 months
  PROMIS-10 Global Health Questionnaire v.1.2 is an NIH-developed, valid and reliable instrument that will be used to assess functional status and quality of life. Higher scores represent better health. Scores will be computed to identify global physical and mental health component scores. Participant patients will complete this assessment at baseline, 2 months, and 5 months (visits 1, 3, and 6, respectively). T-scores will be used in the analysis to identify characteristics associated with other participant patients at the same global health levels. Changes in T-scores over time will be compared with changes in BMI and associated with utilization of the nutrition algorithm.
Symptom Questions | Up to 12 months
  Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAETM) will be used to collect data on the occurrence, severity, and level of interference with daily activities for sleep quality (i.e., insomnia), pain, fatigue, and depression (i.e., anxiety, discouraged, sad) at baseline, 2 months, and 5 months (respectively visits 1, 3, and 6). Higher scores will indicate worse symptom experiences. T-scores will be used in the analysis to identify characteristics associated with other participant patients at the same global health levels. Changes in T-scores over time will be compared with changes in BMI and associated with utilization of the nutrition algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Hammer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT05825469/Prot_SAP_001.pdf